CLINICAL TRIAL: NCT06868043
Title: A Study to Investigate the Function, Safety and Tolerability of a Transdermal Continuous Glucose Monitoring System in Diabetic Patients (Type 1 and 2) for a Period of 28 Days
Brief Title: A Study to Investigate a Transdermal Continuous Glucose Monitoring System in Diabetic Patients for a Period of 28 Days
Acronym: FiberSense
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: One cohort succesfully completed; further cohorts not needed, no safety issue.
Sponsor: EyeSense GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: P-4.2-C-0.1
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Diabetes (DM)
Keywords: diabetes management; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A (Experimental): Subjects will wear 2 FiberSense systems (arm and abdomen) inserted on day 00 and a comparator continuous glucose monitoring (CGM) system on abdomen, changed on weekly basis. They will participate in six clinic in-house sessions on days 00, 03, 07, 14, 21 and 28.
  There will be no home use days, solely several hours of extended use blood glucose readings after selected in-clinic sessions.
  Interventions: Device: FiberSense System
- Cohort B (Experimental): Subjects will wear 2 FiberSense systems (arm and abdomen) inserted on day 00 and a comparator CGM system on abdomen, changed on weekly basis. They will participate in six clinic in-house sessions on days 00, 03, 07, 14, 21 and 28.
  Home use measurement days will be scheduled to wear FiberSense systems for 8-12 hours on days directly before and after a measurement visit day - day 6, 8, 13, 15, 20, 22, and 27.
  Interventions: Device: FiberSense System
- Cohort C (Experimental): Subjects will wear 2 FiberSense systems (arm and abdomen) inserted on day 00 and a comparator CGM system on abdomen, changed on weekly basis. They will participate in six clinic in-house sessions on days 00, 03, 07, 14, 21 and 28.
  Home use measurement days will be scheduled to handle and wear FiberSense systems independently on daily basis (min. 8 hours) between measurement visit days - day 4-6, 8-13, 15-20, and 22-27.
  In addition, interim visits are scheduled at Day 10, 17, and 24 for sensor site and adverse event assessment.
  Interventions: Device: FiberSense System
- Cohort D (Experimental): Subjects will wear 2 FiberSense systems (arm and abdomen) inserted on day 00 and a comparator CGM system on abdomen, changed on weekly basis. They will participate in six clinic in-house sessions on days 00, 03, 07, 14, 21 and 28.
  Home use measurement days will be scheduled to handle and wear FiberSense systems independently on daily basis (min. 8 hours) between measurement visit days - day 4-6, 8-13, 15-20, and 22-27.
  In addition, interim visits are scheduled at Day 10, 17, and 24 for sensor site and adverse event assessment.
  Interventions: Device: FiberSense System

INTERVENTIONS:
Device: FiberSense System — FiberSense system, a novel CGM system using interstitial fluid (ISF) glucose as an indicator of blood glucose levels by diabetic patients

SUMMARY:
Single-centre, open label (unblinded). A maximum of 48 patients will be enrolled in 4 Cohorts of 10 patients and 2 potential replacements each. Diabetic patients (type 1 and 2). Duration up to 11 weeks: up to 6 weeks of screening phase (42 days); 4 weeks of treatment/measurement phase (28 days, depending on sensor functionality) and 1 week of follow up (7 days)

DETAILED DESCRIPTION:
This study is an investigational study, which will be conducted only at one site in Germany. The investigators, the patient and the sponsor will be unblinded.

The eligibility of the patient is determined in up to two steps, a screening (see inclusion criteria) and in case of women of childbearing potential a urine pregnancy test at the day of sensor insertion (independent of any re-screening). Women of childbearing potential are only enrolled after a negative outcome of the urine pregnancy test. The screening results are valid up to 42 days. Within that time the first measurement visit including the insertion of the device should be performed. If the first measurement visit is delayed a re-screening has to be performed. Should the patient not pass the re-screening, the patient is considered as a screening failure and must be excluded.

The trial is structured into three phases, the screening/enrolment phase, the insertion/measurement phase and the follow-up phase.

Screening/Enrolment Phase: Up to 6 weeks (42 days), 1 visit

Insertion/Measurement phase: Up to 4 weeks (28 days), up to 6 in-house measurement visits

Follow-up Phase: 1 week (7 days), 1 visit

ELIGIBILITY:
Inclusion Criteria:

* Body mass index within the range of 19-40 kg/m2, inclusive
* Diabetes type 1 and 2
* Females (if of childbearing potential) must agree to abstain from sexual intercourse or use reliable forms of contraception e.g. condom or diaphragm with spermicide or oral contraceptives to prevent pregnancy during the study
* Negative urine pregnancy test immediately before sensor insertion (only women of childbearing potential)
* Signed written Informed Consent

Exclusion Criteria:

* Inability to follow the protocol schedule
* Participating in another clinical trial
* Pregnant or lactating females, , including positive urine pregnancy test immediately before sensor insertion
* Any known hypersensitivity to any of the products used in the study, including preservatives etc. Especially hypersensitivity against legumes
* Tattoos at the abdominal or upper arm skin area where the fiber sensor is supposed to be placed
* Malignancies requiring therapy during the study
* Severe chronic diseases e.g. renal failure, liver cirrhosis etc. which may interfere with the conduct or completion of the study
* Acute severe infection disease at the time of enrolment
* Alcohol and/or drug addiction
* Vulnerable patients (e.g. persons kept in detention)
* Poorly controlled diabetes mellitus with hemoglobin A1C higher than 10%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Short and mid term performance of the transdermal CGM sensor determined as MARD | 0, 3, 7, 14, 21 and 28 days
  Mean absolute relative difference (MARD) of FiberSense system to blood glucose
Incidence of adverse events | 0, 3, 7,14, 21, 28 and 35-38 days
  Assessment of adverse events and local tolerability occurred during the study

SECONDARY OUTCOMES:
Stability of the blood glucose to fluorescence correlation | 0, 3, 7, 14, 21 and 28 days
  FiberSense fluorescence measurement signals calculated in glucose values and compared to glucose values measured with: a: SMBG device (Bayer Contour next USB), b: CGM device (Dexcom Seven plus), c: Laborat orysystem (Hitado Super GL compact)
Changes in blood glucose to fluorescence lag time over a period of up to 28 days | 0, 3, 7, 14, 21 and 28 days
  Lag time (in minutes) between FiberSense readings and corresponding laboratory blood glucose values during glucose excursions
Correlation between the fluorescence readings of the sensor and capillary blood glucose measurements | 0, 3, 7, 14, 21 and 28 days
  Calculation of MARD of FiberSense against a commercial self-monitoring blood glucose meter
Signal-to-noise ratio | 0, 3, 7, 14, 21 and 28 days
Signal drift | 0, 3, 7, 14, 21 and 28 days
  Drift of the FiberSense fluorescent measurement signals over the wearing time
User satisfaction assessed by the Likert scale | 35-38 days
  Subjective impression of the patients assessed by 5-point Likert scale (1- strongly agree to 5 - strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hasslacher, Prof. Dr., Principal Investigator — Diabetesinstitut Heidelberg
Locations (1):
- Diabetes Instiut Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No